CLINICAL TRIAL: NCT06195306
Title: Phase 2 Study of Low Dose Tamoxifen +/- High Dose Omega-3 Fatty Acids in Overweight Postmenopausal Women at Increased Risk for Breast Cancer
Brief Title: Low Dose Tamoxifen With or Without Omega-3 Fatty Acids for Breast Cancer Risk Reduction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2023-10830; NCI-2023-10830 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UMICC 2024.076 (Other: University of Michigan Rogel Cancer Center); UMI23-14-02 (Other: DCP); P30CA046592 (NIH); UG1CA242632 (NIH)
Record Dates: First submitted 2024-01-04; First posted 2024-01-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Breast Atypical Hyperplasia; Breast Carcinoma; Breast Ductal Carcinoma In Situ; Breast Lobular Carcinoma In Situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Specimen Handling; Omacor; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (tamoxifen) (Experimental): Participants receive tamoxifen PO QD for 180 days in the absence of unacceptable toxicity. Participants may continue to receive tamoxifen PO QD for up to 60 additional days in the case of scheduling delays. Participants also undergo mammography at screening and undergo RPFNA and collection of blood samples at screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Mammography; Other: Questionnaire Administration; Procedure: Random Periareolar Fine-Needle Aspiration; Drug: Tamoxifen
- Group 2 (tamoxifen, omega-3 fatty acids) (Experimental): Participants receive tamoxifen PO QD and omega-3 fatty acids PO BID for 180 days in the absence of unacceptable toxicity. Participants may continue to receive tamoxifen PO QD and omega-3 fatty acids PO BID for up to 60 additional days in the case of scheduling delays. Participants also undergo mammography at screening and undergo RPFNA and collection of blood samples at screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Mammography; Drug: Omega-3-Acid Ethyl Esters; Other: Questionnaire Administration; Procedure: Random Periareolar Fine-Needle Aspiration; Drug: Tamoxifen

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Mammography — Undergo mammography
  Other Names: MG
Drug: Omega-3-Acid Ethyl Esters — Given PO
  Other Names: Lovaza
  Arms: Group 2 (tamoxifen, omega-3 fatty acids)
Other: Questionnaire Administration — Ancillary studies
Procedure: Random Periareolar Fine-Needle Aspiration — Undergo RPFNA
  Other Names: Random Periareolar Fine Needle Aspiration; RPFNA
Drug: Tamoxifen — Given PO
  Other Names: TMX

SUMMARY:
This phase II trial evaluates tamoxifen, with or without omega-3 fatty acids, for reducing risk of breast cancer among postmenopausal and overweight or obese women who are at increased risk of developing breast cancer. Tamoxifen is a selective estrogen receptor modulator. It works by blocking the effects of the hormone estrogen in the breast. Tamoxifen is approved by the Food and Drug Administration for prevention of breast cancer in women at increased risk. Omega-3 fatty acids have been shown to decrease the amount of fats made in the liver. Omega-3 fatty acids may work to prevent cancer in overweight or obese individuals. Tamoxifen with or without omega-3 fatty acids may be effective at reducing risk of breast cancer among women who are postmenopausal, overweight or obese, and at increased risk.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate average change in serum adiponectin within the low dose tamoxifen (LDTAM) + high dose omega-3-acid ethyl esters (omega-3 fatty acids) arm.

II. To study the beneficial effects of addition of high dose omega-3 fatty acids to LDTAM by comparing the relative difference in change in serum adiponectin in overweight and obese high-risk postmenopausal women randomized to 6 months of LDTAM or LDTAM + high dose omega-3 fatty acids.

SECONDARY OBJECTIVES:

I. To determine effect of LDTAM +/- high dose omega-3 fatty acids on insulin resistance, insulin sensitivity, and insulin secretory function (homeostatic model assessment for insulin resistance [HOMA-IR], homeostatic model assessment of insulin sensitivity [HOMA%S] homeostatic model assessment of beta cell function, [HOMA%B]), respectively.

II. To determine effect of LDTAM +/- high dose omega-3 fatty acid on benign breast tissue estrogen response gene index (ERGI).

EXPLANATORY OBJECTIVES:

I. Effect of change in red blood cell (RBC) omega-3:omega-6 fatty acid ratio on within arm change in blood adiponectin.

II. Effect of change in RBC omega-3:omega-6 fatty acid ratio on within arm change in tissue ERGI.

III. Effect of baseline bioavailable estradiol on within arm change in blood adiponectin.

IV. Effect of baseline and 6-month bioavailable estradiol on within arm change in tissue ERGI.

V. Effect of 6-month tamoxifen active metabolites (endoxifen and 4-hydroxy [4OH] tamoxifen) on change in ERGI.

VI. Effect of eicosapentaenoic acid/docosahexaenoic acid (EPA/DHA) dietary intake as measured by DHA Food Frequency Questionnaire on RBC omega 3:6 fatty acid ratio change.

EXPLORATORY OBJECTIVES:

I. Assess within arm effects of LDTAM +/- high dose omega-3 fatty acids on serum triglycerides.

II. Assess within arm effects of LDTAM +/- high dose omega-3 fatty acids on adiponectin:leptin ratio.

III. Assess within arm effects of LDTAM +/- high dose omega-3 fatty acids on anterior gradient protein 2 homolog (AGR2) messenger ribonucleic acid (mRNA).

IV. Assess within effects of LDTAM +/- high dose omega-3 fatty acids on forkhead box A1 (FOXA1) protein (immunohistochemistry [IHC]).

V. Assess within arm effects of LDTAM +/- high dose omega-3 fatty acids on AGR2 protein (IHC).

VI. Assess effects of LDTAM +/- high dose omega-3 fatty acids on Ki-67 (IHC) in individuals with > 500 cells in baseline ThinPrep and measurable baseline Ki-67.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP 1: Participants receive tamoxifen by mouth (PO) once daily (QD) for 180 days in the absence of unacceptable toxicity. Participants may continue to receive tamoxifen PO QD for up to 60 additional days in the case of scheduling delays. Participants also undergo mammography at screening and undergo random periareolar fine needle aspiration (RPFNA) and collection of blood samples at screening and on study.

GROUP 2: Participants receive tamoxifen PO QD and omega-3 fatty acids PO twice daily (BID) for 180 days in the absence of unacceptable toxicity. Participants may continue to receive tamoxifen PO QD and omega-3 fatty acids PO BID for up to 60 additional days in the case of scheduling delays. Participants also undergo mammography at screening and undergo RPFNA and collection of blood samples at screening and on study.

After completion of study intervention, participants are followed up at 21-35 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 - 65
* Postmenopausal female

  * Postmenopausal is defined as either

    * Prior removal of the ovaries, or if ovaries intact amenorrhea for >= 12 months and not on any form of contraception, or
    * Amenorrhea for greater than 2 months with serum follicle-stimulating hormone (FSH) in postmenopausal range (>= 25 IU/L). Women with ovaries and a prior hysterectomy or endometrial ablation < age 55 must have a FSH >= 25 IU/L. Women may be on vaginal low dose estrogen preparations for vaginal dryness. Women over age 50 with a levonorgestrel intrauterine device in place for 2 or more years and not planning removal in the next 6 month are also eligible if FSH >= 25 IU/L

      * Note: FSH will be done at time of screening
* Women with intact ovaries and uterus < age 55 must have a negative pregnancy test prior to randomization
* Overweight or obese (body mass index [BMI] >= 25 kg/m^2)

  * Note: BMI must be calculated within 28 days of randomization
* Willing to undergo a fasting blood draw and non-fasting RPFNA with fixed and frozen aliquots sent to University of Kansas Medical Center (KUMC)
* At increased risk of breast cancer per at least one of the following:

  * Personal medical history

    * History of atypical hyperplasia or lobular carcinoma in situ (LCIS) found on breast biopsy
    * History of unilateral ductal carcinoma in situ treated with unilateral mastectomy, lumpectomy, or local excision with or without radiation and this treatment was completed at least 3 months prior to the screening RPFNA
    * High mammographic density determined by one of the following:

      * Visual estimate of area of density (VAS) > 50%,
      * Volpara (trademark) >= 15% dense volume (Volpara d)
      * Breast Imaging Reporting and Data System (BIRADS) assessment = extremely dense (BIRADs D)
  * Genetic test result

    * Germline gene mutation in ATM, BARD1, BRCA2, CDH1, CHEK2, NF1, PALB2, PTEN, RAD51C, RAD51D, or STK11
    * Polygenic lifetime risk score >= 2x average or 25%
  * Calculated risk based on standard models

    * Five-year Breast Cancer Risk Assessment Tool (BCRAT) (version 2.0) >= 1.66%
    * Ten-year International Breast Cancer Intervention Study risk evaluation tool (IBIS) (version 8) >= 3%
    * Ten-year relative risk IBIS (version 8) >= 2X that for age group
    * Ten- year Breast Cancer Surveillance Consortium (version 2) >= 3%
  * Family History

    * Breast cancer in a first or second degree relative (female or male) with onset under age 50. (First degree relative = parent, sibling, or child. Second degree relative = grandparent, uncle, aunt, nephew, niece, half-sibling, grandchild or first cousin)
    * Breast cancer in two or more first or second-degree relatives from either the maternal or paternal linage without regard to age
    * Bilateral breast cancer or breast and ovarian cancer in the same first or second degree relative without regard to age
  * Primary source documentation of risk is required and must be submitted to the lead academic organization (LAO) for review along with the eligibility checklist

    * Risk factor: Atypical hyperplasia or LCIS; Primary source document: Copy of pathology report or clinical note confirming the diagnosis
    * Risk factor: Ductal carcinoma in situ (DCIS) and treatment history; Primary source document: Copies of pathology report or clinic notes confirming the diagnosis, treatment plan and treatment end date(s)
    * Risk factor: Mammographic density; Primary source document: Copy of clinic note or mammogram report
    * Risk factor: Genetic; Primary source document: Copy of genetic test report
    * Risk factor: Calculated based on standard models; Primary source document: Copy of the calculation result
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)

  * Note: Higher total bilirubin levels (=< 3 mg/dL) can be allowed if due to known benign liver condition, i.e., Gilbert's syndrome
  * Results from prior laboratory testing within 180 days of randomization may be used
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) =< 3.0 x institutional upper limit of normal

  * Results from prior laboratory testing within 180 days of randomization may be used
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional upper limit of normal

  * Results from prior laboratory testing within 180 days of randomization may be used
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients on chronic suppressive antiviral therapy for herpes simplex virus (HSV) are eligible
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Women must have at least 1 unaffected untreated breast for fine needle aspiration. Women may have had prior unilateral breast radiation or mastectomy for DCIS
* Ability to understand and the willingness to sign a written informed consent document
* Most recent screening mammogram must be performed ≤ 12 months prior to RPFNA and must be reported as BIRAD 1 or 2. If BIRAD 0 then follow-up diagnostic imaging must be BIRAD 1 or 2 or cleared clinically with radiology recommendation of return to annual screening
* Confirmation that baseline research blood was drawn fasting (>= 10 hours), has been received in good condition at KUMC, and is archived for assessment of primary endpoint

Exclusion Criteria:

* Exclusions based on current or past conditions:

  * Bilateral breast implants (danger of implant puncture with RPFNA)
  * Prior invasive breast cancer
  * Prior invasive uterine cancer
  * Other prior invasive cancer and haven't completed cancer related therapy or with evidence of disease (other than non-melanoma skin cancer) within the past 2 years
  * Currently breastfeeding (concern that tamoxifen may be in breast milk) or nursing within past 12 months (concern about milk fistula with RPFNA)
  * Type I or type II diabetes mellitus requiring current pharmacologic treatment (including metformin, glucagon-like peptide 1 agonists, insulin, sulfonylurea)
  * Prior deep vein thrombosis, pulmonary embolus, or stroke
  * Prior gastric bypass surgery
  * History of chronic liver disease including NASH (nonalcoholic steatohepatitis) or cirrhosis
  * Pathogenic or likely pathogenic germline mutation in BRCA1 or TP53
* Exclusions based on medications:

  * Current use of prescription anticoagulants such as Coumadin (warfarin), direct-acting oral anticoagulants such as Xarelto (rivaroxaban) or Eliquis (apixaban) or heparin
  * Women who would not be able to or do not wish to discontinue daily use of aspirin (81mg or higher) and aspirin containing products (81 mg or higher) at least 3 weeks prior to each RPFNA

    * Note: Women may resume daily use of aspirin and aspirin containing products 3 days after each RPFNA procedure
  * Current use of a levonorgestrel intrauterine device if in place less than 2 years or if there is planned removal within the next 6 months
  * Current use of hormone therapy (oral, transdermal, or injectable)

    * Note: Vaginal estrogen is allowed
  * Prior treatment with tamoxifen, aromatase inhibitor or selective estrogen receptor degrader for more than 2 months

    * Note: Women with < 2 months of these drugs must be off for at least 6 months before they may begin biomarker screening tests
  * Greater than 1 gram daily of omega-3 fatty acid supplement within the last 6 months
  * Current use of prescription immunosuppressive drugs
  * Current use of CYP3A4 strong inducers rifampin or aminoglutethimide
  * Current use of or plans to initiate a glucagon-like peptide 1 agonist within the next 6 months
  * Current use of metformin for any indication
* Participants may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to tamoxifen or omega-3 fatty acid or generic Lovaza or compounds of similar chemical composition
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in serum adiponectin | From baseline up to end of treatment (6 months)
  An analysis for difference between the two arms will be conducted to document a beneficial effect of addition of high dose omega-3 fatty acids to low dose tamoxifen. Paired and unpaired t-tests will be used.

SECONDARY OUTCOMES:
Change in insulin resistance | From baseline up to end of treatment (6 months)
  Evaluated using Homeostatic Model Assessment of Insulin Resistance, as calculated using fasting glucose and fasting insulin. Paired and unpaired t-tests will be used. Spearman correlation between change in biomarkers will be estimated and compared across the study arms using Fisher's Z-transformed values.
Change in insulin sensitivity | From baseline up to end of treatment (6 months)
  Evaluated using Homeostatic Model Assessment of Insulin Sensitivity. Paired and unpaired t-tests will be used. Spearman correlation between change in biomarkers will be estimated and compared across the study arms using Fisher's Z-transformed values.
Change in insulin secretory function | From baseline up to end of treatment (6 months)
  Evaluated using Homeostatic Model Assessment of Beta Cell Function. Paired and unpaired t-tests will be used. Spearman correlation between change in biomarkers will be estimated and compared across the study arms using Fisher's Z-transformed values.
Estrogen response gene index (ERGI) | From baseline up to end of treatment (6 months)
  The estrogen response gene index reflects change in gene expression over time. The genes assayed for this index are: ESR1 (codes for estrogen receptor alpha), ESR2 (codes for estrogen receptor beta), GREB1 (codes for growth regulation by estrogen in breast cancer 1), PGR (codes for progesterone receptor) and TFF1 (also known as pS2, which codes for trefoil factor 1). The log2-transformed values of the ratio of relative abundance (6-month value: baseline value) for GREB1, PGR, TFF1, and the ratio of ESR1:ESR2 are averaged to produce the ERGI. Paired and unpaired t-tests will be used. Spearman correlation between change in biomarkers will be estimated and compared across the study arms using Fisher's Z-transformed values.

OTHER OUTCOMES:
Effect of change in red blood cell omega-3:omega-6 fatty acid ratio on within arm change in blood adiponectin | Up to 6 months
Effect of change in red blood cell omega-3:omega-6 fatty acid ratio on within arm change in tissue ERGI | Up to 6 months
Effect of baseline bioavailable estradiol on within arm change in blood adiponectin | Up to 6 months
Effect of baseline and 6-month bioavailable estradiol on within arm change in tissue ERGI | Up to 6 months
Effect of 6-month tamoxifen active metabolites on change in ERGI | Up to 6 months
Effect of eicosapentaenoic acid/docosahexaenoic acid dietary intake on red blood cell omega-3:omega-6 fatty acid ratio change | Up to 6 months
Serum triglycerides | Up to 6 months
  Will evaluate within arm effects of low dose tamoxifen +/- high dose omega-3 fatty acids on this exploratory outcome.
Adiponectin:leptin ratio | Up to 6 months
  Will evaluate within arm effects of low dose tamoxifen +/- high dose omega-3 fatty acids on this exploratory outcome.
Anterior gradient protein 2 homolog messenger ribonucleic acid | Up to 6 months
  Will evaluate within arm effects of low dose tamoxifen +/- high dose omega-3 fatty acids on this exploratory outcome.
Forkhead box A1 protein | Up to 6 months
  Will evaluate within arm effects of low dose tamoxifen +/- high dose omega-3 fatty acids on this exploratory outcome.
Anterior gradient protein 2 homolog protein | Up to 6 months
  Will evaluate within arm effects of low dose tamoxifen +/- high dose omega-3 fatty acids on this exploratory outcome.
Ki-67 | Up to 6 months
  Will evaluate within arm effects of low dose tamoxifen +/- high dose omega-3 fatty acids on this exploratory outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Nye, Principal Investigator — University of Kansas
Locations (3):
- United States (3):
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm